CLINICAL TRIAL: NCT06273904
Title: Modulating Escape in the Anxiety Disorder Spectrum: Targeting the Direct Neural Mediator Using Transcranial Focused Ultrasound
Brief Title: Modulating Escape Using Focused Ultrasound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Christopher Sege, Research Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00132631
Record Dates: First submitted 2024-02-13; First posted 2024-02-23 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Group Receiving Active Stimulation and Sham Stimulation on Separate Days (All Participants) (Experimental): All participants will receive active stimulation and non-active (sham) stimulation on different days. Before the stimulation sessions, all participants will complete experimental tasks during functional magnetic resonance imaging. On the next two study days, all participants will complete tasks before and after receiving active transcranial focused ultrasound (tFUS) on one day and sham (non-active) tFUS on another day. Stimulation (active or sham) is conducted briefly (< 10 minutes) in between tasks, not during tasks.
  Interventions: Device: Active transcranial focused ultrasound (tFUS); Device: Sham transcranial focused ultrasound (tFUS)

INTERVENTIONS:
Device: Active transcranial focused ultrasound (tFUS) — Active non-invasive low-intensity focused ultrasound will be delivered using a proprietary head-worn device and control software from Attune Neurosciences. On an active stimulation day, focused ultrasound will be delivered to the brain region of interest using parameters from published research that are demonstrated to safely cause temporary changes in the activity in that brain area.
Device: Sham transcranial focused ultrasound (tFUS) — Non-active low-intensity ultrasound will also be conducted using a proprietary head-worn device and control software from Attune Neurosciences. On the sham stimulation day, the device will be activated in a manner that produces similar sensory effects (i.e., low-volume beeping-type noise from the device) but also prevents delivery of a focused ultrasound beam to the brain area of interest or any other brain area.

SUMMARY:
This is a study to find out if a cutting-edge technology called transcranial focused ultrasound (tFUS) can be used to treat how people with anxiety or related concerns cope with emotional situations. tFUS is a brain stimulation technology that causes temporary changes in the activity of deep brain areas without a need for any surgery or other permanent or invasive procedures.

This study is recruiting participants who recently started treatment for anxiety or a related concern to come in for 3 visits at the Medical University of South Carolina. At the first visit, participants will do interviews and surveys asking about anxiety and related concerns, and they do tasks where they respond to emotional pictures while brain activity is measured using magnetic resonance imaging (MRI). At the next two visits, participants again do a task where they see and react to emotional images, and this time the task is done once before and again once after receiving tFUS that either actively causes temporary changes (lasting for about an hour) in a targeted brain area or is not active (no changes elicited). At each tFUS visit, responses are measured with sensors worn on the hand, arms, face, and head (these visits do not involve MRI).

Each visit in this study is expected to last between 2 - 3 hours. This study is not a treatment study, but it could help improve treatment in the future. Participants in this study are paid for their time.

DETAILED DESCRIPTION:
Escape and avoidance are core targets of anxiety and related disorder treatment, but such behaviors also often persist even after reduction of reported symptoms or they keep an individual from engaging in treatment at all. Novel methods to directly target motive drivers of escape/ avoidance coping early in treatment are needed to improve retention and outcome especially for the 20% of individuals who do not benefit from and 40% who do not complete treatment. Basic science identifies multiple neural mediators of real-world escape and avoidance, and it suggests these mediators may not be directly or adequately targeted by current treatment techniques. Moreover, the direct neural mediators may be primarily subcortical and thus not be accessible to therapeutic technologies like transcranial magnetic stimulation that can only stimulate cortical areas. A novel technology called transcranial focused ultrasound (tFUS), meanwhile, has demonstrated ability to non-invasively and stimulate even the deepest areas of the brain in humans, and thus may have utility in directly modulating the subcortical drivers of exaggerated escape/ avoidance coping. Given this exciting possibility, the primary goal of this research is to determine if tFUS to subcortical neural mediators can be used to cause measurable changes in the downstream escape/ avoidance dispositions. Results will then inform the potential use of noninvasive tFUS stimulation as a precursor to evidence-based therapy to reduce risk of dropout and enhance outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 y.o.
* Meets criteria for an anxiety disorder (Generalized Anxiety Disorder, Panic Disorder, Social Anxiety Disorder, Specific Phobia), posttraumatic stress disorder, obsessive-compulsive disorder, or current adjustment disorder with anxiety
* Is currently seeking mental health treatment
* Is able to read consent document and provide informed consent.
* English is a first or primary fluent language.

Exclusion Criteria:

* Current alcohol or substance use disorder of more than mild severity (as defined by the Diagnostic and Statistical Manual (DSM)-5 and determined using standardized self-report instruments)
* Lifetime diagnosis of psychotic disorder or bipolar mania
* Presence of neurological disorder that contraindicates brain stimulation or neurophysiological recording: Seizure disorder
* Lifetime history of traumatic brain injury with loss of consciousness
* Neurodegenerative disorder (e.g., Alzheimer's Disease, Parkinson's Disease, Frontotemporal Dementia)
* Presence of other medical disorder that would make it too uncomfortable to sit or lie still for long recording periods
* Presence of standard contraindications for magnetic resonance imaging
* Metal in the body
* Currently pregnant
* Claustrophobia
* Significant sensitivity to noise
* Medical conditions or treatments that lower seizure threshold
* History of severe brain injury
* History of seizures/ epilepsy
* Currently taking anticholinergic mediation, neuroleptic medication, or sedative/ hypnotic medication

Note: selective serotonin re-uptake inhibitors (SSRIs), cholinesterase inhibitors or N-methyl-D-aspartate (NMDA) receptor antagonists are allowed if patient has been on a stable regimen of four weeks prior to enrollment

* Currently taking chronic opiate medications or substances
* Currently taking naltrexone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Fear-Potentiated Startle Reflex | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 10 minutes between assessments)
  Fear-potentiated startle is measured during an experimental task in which participants prepare to avoid, escape, or simply be exposed to aversive pictures. Fear-potentiated startle measures motivational activation during the preparation period.

SECONDARY OUTCOMES:
Change in speed to initiate avoidance behavior | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 10 minutes between assessments)
  Reaction time to initiate flight is measured in an experimental task in which participants change the size of pleasant or unpleasant images with a joystick. Reaction time measures behavioral tendency toward avoidance in the presence of unpleasant images or approach in the presence of pleasant images
Change in Electroencephalography (EEG)-Assessed Contingent Negative Variation During Escape/ Avoidance Preparation | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 10 minutes between assessments)
  Brain electroencephalography (EEG) is measured non-invasively with sensors placed on top of the head during all pre/ post-stimulation experimental tasks. The Contingent Negative Variation (CNV) is an event-related potential measure of motor preparation processing that arises in S1-S2-type tasks.
Change in Electroencephalography (EEG)-Assessed N200 During Implicit Approach/ Avoid Bias Assessment | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 10 minutes between assessments)
  Brain electroencephalography (EEG) is measured non-invasively with sensors placed on top of the head during all pre/ post-stimulation experimental tasks. The N200 is an event-related potential measure of neural stimulus-response conflict that can be used to index the degree to which unpleasant stimuli facilitate avoidant behavior.
Change in Electroencephalography (EEG)-Assessed Theta-Band Power During Behavioral Tasks | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 10 minutes between assessments)
  Brain electroencephalography (EEG) is measured non-invasively with sensors placed on top of the head during all pre/ post-stimulation experimental tasks. Power in a theta frequency band is a measure of cognitive control that will be assayed in all behavioral tasks as a measure of task engagement changes
Change in High-Frequency Heart Rate Variability/ Respiratory Sinus Arrhythmia | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 10 minutes between assessments)
  Heart rate and also respiration are measured during all pre/ post-stimulation experimental tasks. These measures can be combined to derive an index of the strength of vagal control over the heart (High-Frequency Heart Rate Variability/ Respiratory Sinus Arrhythmia) that reflects greater attentional control relative to stress (i.e., sympathetic) responding. This measure will be assayed in all tasks and in resting measurements conducted pre- and post-stimulation.
Change in Task-Based Heart Rate (Beats per Minute) Changes | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 10 minutes between assessments)
  Heart rate is measured during all pre/ post-stimulation experimental tasks. Task event-related changes in heart rate will be measured as an index of the strength of attentional orienting to all motivationally relevant cues
Change in Task-Based Galvanic Skin Conductance | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 10 minutes between assessments)
  Skin conductance is measured during all pre/ post-stimulation experimental tasks from sensors placed on the hand. Skin conductance can be indexed to test for changes in sympathetic activation during escape/ avoidance preparation.
Change in State Anxiety During Session | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 10 minutes between assessments)
  State-level anxiety is measured throughout the experimental session using the State-Trait Anxiety Inventory - State Form. The State-Trait Anxiety Inventory - State Form uses 20 items querying anxiety symptom experience in the present moment to measure how anxiety fluctuates across the experimental session. The scale ranges from 20 to 80, with higher scores indicating higher state anxiety.

OTHER OUTCOMES:
Task-Related Regional Brain Activation | During Session (Approx. 45 minutes)
  Blood flow in the brain will be measured during completion of an experimental escape/ avoidance task using functional magnetic resonance imaging (fMRI). Blood flow in the brain can be used to measure what brain areas are being activated during the performance of a task.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sege, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No